CLINICAL TRIAL: NCT02506543
Title: Creating Opportunities Through Mentoring, Parental Involvement and Safe Spaces - Ethiopia
Acronym: COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: International Rescue Committee (Other); Department for International Development, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Lindsay Stark, Associate Professor of Population and Family Health at the Colum, Dept Population&Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAP6855
Record Dates: First submitted 2015-07-19; First posted 2015-07-23 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Sexual Assault; Interpersonal Relations; Marital Status; Domestic Violence
Keywords: Adolescent Health; Ethiopia; Sexual Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COMPASS intervention (Experimental): Subjects in this group will be pre-tested at the same time with the subjects in the Wait-list control group. Subjects in this group will receive the intervention immediately after the initial pre-test/baseline assessment, which includes life skills education, access to mentors in safe spaces, and a structured parenting intervention for girls' caregivers. Then, the subjects in this group have completed the intervention (at 12-months post-intervention initiation), the subjects in this group will take the post-test at the same time with the subjects in the Wait-list control group.
  Interventions: Behavioral: COMPASS
- Wait-list control (Active Comparator): No intervention
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: COMPASS — COMPASS (Creating Opportunities through Mentoring, Parental involvement and Safe Spaces) is a program for 13-19 year old girls in three refugee camps in Ethiopia. The program is a structured intervention that is intended to engage adolescent girls, through life skills training and establishing or supporting community-supported safe spaces for girls where they can come and gather among themselves and participate in a structured life-skills curriculum.
  Arms: COMPASS intervention
Behavioral: No intervention — Wait list control group will not receive an intervention. After the follow-up study, the wait-list control group will receive the regular COMPASS program
  Arms: Wait-list control

SUMMARY:
The study is a randomized controlled trial of COMPASS, an intervention for adolescent girls in three refugee camps in Ethiopia. The study design will employ a two group wait-list cluster randomized controlled trial where girls will be invited to participate in the COMPASS program, assigned to groups of approximately 20 for the purposes of the program, complete a pre-test baseline assessment, and will then be randomized by group to the intervention or control condition. In addition, qualitative research will address additional questions of acceptability, processes of change and best practice.

Groups in three refugee camps - Sherkole, Bambasi, and Tongo - will be randomized to determine whether the participants receive the intervention or are placed on the wait-list immediately following the baseline. Those that do not get the curriculum during the study will receive it following the endline phase of the study so as to not create tensions or jealousies.

The intervention, the COMPASS program, will involve a structured intervention for girls between the ages of 13-19 that is intended to engage adolescent girls, those who are influential in their lives, service providers and other stakeholders, with the ultimate goal of co-creating environments in which girls are valued and safe. The program is centered on establishing or supporting community-supported safe spaces for girls where they can come and gather among themselves and participate in a structured life-skills curriculum.

DETAILED DESCRIPTION:
The study assessment will employ a mixed methods approach with most data collection occurring at pre-test/baseline and post-intervention. Quantitative survey methods will be used to evaluate attitudes towards a host of topics related to physical and financial assets and health-related behaviors. Survey questions will be administered using Audio Computer Assisted Self-Interviewing (ACASI). Quantitative methods will be used to yield statistical measures of the scale of changes in attitudes, skills, and behaviors due to the intervention.

Qualitative methods at baseline will include focus group discussions with caregivers and participatory methods with girls to assess topics such as self-esteem, empowerment, safety, and resilience. Endline qualitative methods include in-depth interviews with caregivers, and small-group warm-up activities with adolescent girls, followed by in-depth interviews.

ELIGIBILITY:
Inclusion Criteria:

* female
* aged 13-19
* speak one of the languages included in the study (Sudanese Arabic, Funj/Berta, Maban, Regarig and Engesena Quickly dialects)
* give informed consent

Exclusion Criteria:

* cognitive impairment

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1014 (Actual)
Dates: Start 2015-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Sexual violence in the past 12 months | 12 months
  A binary composite representing any form of sexual violence in the previous 12 months, which included self-reported forced sex, unwanted sexual touching, or coerced sex

SECONDARY OUTCOMES:
Change in baseline prevalence of interpersonal relationships | 12 months
  This study will use a questionnaire to measure whether there is an increase in study participants' average number close friends from the pre-test to post-test evaluation. Girls will also self-report sources of emotional support such as comfort in discussing problems with a trusted female adult and comfort discussing topics such as education, marriage, puberty, pregnancy prevention, HIV/AIDS, and financial plans with caregivers.
Change in baseline prevalence of physical abuse | 12 months
  This study will use a questionnaire to measure whether the percentage of girls who self-reported experiencing beatings within the past 12 months decreases between the pre-test and post-test evaluation.
Change in baseline prevalence of early marriage | 12 months
  This study will use a questionnaire to measure changes in the percentage of girls who self-reported being married from the pre-test to post-test evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Stark, PhD, Principal Investigator — Associate Professor of Population and Family Health, Columbia University
Locations (2):
- Columbia University, New York, New York, United States
- International Rescue Committee, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stark L, Asghar K, Seff I, Yu G, Tesfay Gessesse T, Ward L, Assazenew Baysa A, Neiman A, Falb KL. Preventing violence against refugee adolescent girls: findings from a cluster randomised controlled trial in Ethiopia. BMJ Glob Health. 2018 Oct 19;3(5):e000825. doi: 10.1136/bmjgh-2018-000825. eCollection 2018. PMID 30398223
- [Derived] Falb KL, Tanner S, Ward L, Erksine D, Noble E, Assazenew A, Bakomere T, Graybill E, Lowry C, Mallinga P, Neiman A, Poulton C, Robinette K, Sommer M, Stark L. Creating opportunities through mentorship, parental involvement, and safe spaces (COMPASS) program: multi-country study protocol to protect girls from violence in humanitarian settings. BMC Public Health. 2016 Mar 5;16:231. doi: 10.1186/s12889-016-2894-3. PMID 26945586